CLINICAL TRIAL: NCT00979992
Title: A Phase II Evaluation of SU11248 (Sunitinib Malate) (NSC #736511) in the Treatment of Persistent or Recurrent Clear Cell Ovarian Carcinoma
Brief Title: Sunitinib Malate in Treating Patients With Persistent or Recurrent Clear Cell Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-03811; NCI-2011-03811 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000654556; GOG-0254 (Other: NRG Oncology); GOG-0254 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Ovarian Clear Cell Adenocarcinoma; Recurrent Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (sunitinib malate) (Experimental): Patients receive sunitinib malate PO QD for 4 weeks. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Sunitinib Malate

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Sunitinib Malate — Given PO
  Other Names: SU011248; SU11248; sunitinib; Sutent

SUMMARY:
This phase II trial studies the side effects of sunitinib malate and how well it works in treating patients with ovarian cancer that is persistent or has come back. Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the anti-tumor activity of SU11248 (sunitinib malate), a highly potent, selective tyrosine kinases inhibitor, in patients with persistent or recurrent clear cell ovarian carcinoma.

II. To examine the nature and degree of toxicity in this cohort of patients treated with this regimen.

SECONDARY OBJECTIVES:

I. To characterize the distribution of progression-free survival and overall survival for patients treated with SU11248 (sunitinib malate).

TERTIARY OBJECTIVES:

I. To determine the pre-cycle 1, pre-cycle 4 and off-treatment levels of pro-angiogenic proteins (e.g., angiogenin, soluble vascular cell adhesion molecule [VCAM]-I, basic fibroblast growth factor [bFGF], platelet-derived growth factor [PDGF], placental growth factor [PlGF], vascular endothelial growth factor [VEGF], and hypoxia-inducible factor [HIF]1alpha).

II. To identify changes in serum and plasma angiogenesis markers at baseline (pre-cycle 1), during treatment (cycle 4), and at progression in association with primary and secondary clinical endpoints associated with clinical response or progression-free survival.

OUTLINE:

Patients receive sunitinib malate orally (PO) once daily (QD) for 4 weeks. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent clear cell ovarian cancer; primary tumors must be at least 50% clear cell histomorphology in order to be eligible or have a histologically documented recurrence with at least 50% clear cell histomorphology; in addition, the tumors should be negative for expression of Wilms tumor (WT)-1 antigen and estrogen receptor (ER) antigen by immunohistochemistry; appropriate tissue sections must be available for histologic evaluation for central pathology review by Gynecologic Oncology Group (GOG); immunohistochemical stained slides for ER and WT-1 antigen must be available for review by GOG

  * If the primary tumor had at least 50% clear cell histomorphology, a biopsy of the recurrent or persistent tumor is not required; however, immunohistochemical studies of the primary tumor for ER and WT-1 antigens should be performed and the slides submitted to the GOG for review; the percentage of clear cell histomorphology must be documented in the pathology report or in an addendum to the original report; if slides of the primary tumor are not available for review due to disposal of slides by the histology laboratory (typically 10 years after diagnosis), biopsy of recurrent or persistent disease is required
  * If the primary tumor had less than 50% clear cell histomorphology (or if slides of the primary tumor are not available for review), a biopsy of the recurrent or persistent tumor is required to confirm at least 50% clear cell histomorphology and lack of immunoreactivity for ER and WT-1 antigens by immunohistochemistry; the percentage of involvement must be documented in the pathology report or in an addendum to the original report
* All patients must have measurable disease as defined by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patients must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy; thus, a confirmed biopsy in an irradiated area at a date longer than 90 days post-completion of radiation can be considered a target lesion to assess progression and response
* Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound; this initial treatment may have included intraperitoneal therapy, consolidation, or extended therapy administered after surgical or non-surgical assessment
* Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of recurrent or persistent disease according to the following definition:

  * Cytotoxic regimens include any agent that targets the genetic and/or mitotic apparatus of dividing cells, resulting in dose-limiting toxicity to the bone marrow and/or gastrointestinal mucosa
* Patients who have received only one prior cytotoxic regimen (platinum-based regimen for management of primary disease) must have a platinum-free interval of less than 12 months, or have progressed during platinum-based therapy, or have persistent disease after a platinum-based therapy
* Patients may have received prior biologic therapy, but must not have had any prior therapy with agents which inhibit VEGF, vascular endothelial growth factor receptor (VEGFR) or PDGF such as, bevacizumab, sorafenib, sunitinib, pazopanib, brivanib, aflibercept cediranib, BIBF 1120, imatinib, dasatinib
* Any other prior therapy directed at the malignant tumor, including immunologic agents (e.g. tamoxifen) must be discontinued at least three weeks prior to registration
* Patients must not be eligible for a higher priority (e.g.; Phase III), GOG protocol for the same population if one exists
* Patients must be recovered from effects of recent surgery (28 days must elapse between surgery and the start of treatment with sunitinib malate)
* Patents must have >= 4 weeks since prior chemotherapy or radiation (>= 6 weeks for nitrosoureas or mitomycin C)
* Sunitinib metabolizes via liver enzyme, specifically the cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) enzyme; therefore, potential drug interaction with the CYP3A4 enzyme can occur; eligible patients who are on the CYP3A4 inducer or inhibitor enzyme should stop 2 weeks prior to study entry if all other eligibility has been confirmed; the principal investigator will review the case and make all effort to switch such agent to other medication
* Patients should be free of active infection (with the exception of uncomplicated urinary tract infections [UTI]) requiring antibiotics
* Patients who have received one prior regimen must have a GOG performance status of 0, 1 or 2; patients who have received two prior regimens must have GOG performance status of 0 or 1
* Absolute neutrophil count (ANC) >= 1,500/mcl
* Platelets greater than or equal 100,000/mcl
* Creatinine less than or equal to 1.5 times the upper limit of normal (ULN)
* Bilirubin less than or equal to 1.5 ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 2.5 times the ULN, unless subjects have liver metastasis, in which case both AST and ALT must be less than or equal to 5 times the ULN
* Patients who have met the pre-entry requirements
* Patients must have signed an approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* Primary peritoneal or fallopian tube primaries are not eligible
* Patients with serious non-healing wound, ulcer, or bone fracture
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels
* Patients with history or evidence upon physical examination of central nervous system (CNS) disease, including primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of cerebrovascular accident (CVA, stroke), transient ischemic attack (TIA) or subarachnoid hemorrhage within 6months of the first date of treatment on this study
* Patients with clinically significant cardiovascular disease; this includes:

  * Poorly controlled hypertension (systolic blood pressure of >= 140 mm Hg or diastolic blood pressure of >= 90 mm Hg) are ineligible
  * Myocardial infarction or unstable angina within 6 months prior to registration
  * New York Heart Association (NYHA) grade II or greater congestive heart failure
  * Cardiac arrhythmia requiring medication
  * Grade II or greater peripheral vascular disease based on National Cancer Institute Common Terminology Criteria (NCI CTC); e.g. ischemic rest pain, minor tissue loss, and ulceration or gangrene
* Patients with QTc prolongation (> 500 msec) are excluded
* Patients who require use of therapeutic doses of Coumadin-derivative anticoagulants such as warfarin are ineligible, although doses of up to 2 mg daily are permitted for prophylaxis of thrombosis; low molecular weight heparin is permitted provided patient's prothrombin time (PT) international normalized ratio (INR) is =< 1.5
* Patients with clinically significant peripheral artery disease, e.g., those with claudication, within 6 months
* Patients with a pre-existing thyroid abnormality who are unable to maintain thyroid function in the normal range with medication are ineligible; patients with a history of hypothyroidism are eligible provided they are currently euthyroid
* Patients whose circumstances do not permit completion of the study or the required follow-up
* Patients who are pregnant or nursing; to date, no fetal studies in animals or humans have been performed; the possibility of harm to a fetus is likely; this drug specifically inhibits VEGF, which is responsible for formation of new blood vessels during development, and antibodies can cross the placenta; therefore, it should not be administered to pregnant women; subjects will be apprised of the large potential risk to a developing fetus; it is not known whether the drug is excreted in human milk; because many drugs are excreted in human milk, this drug should not be administered to nursing women; women of childbearing potential must agree to use contraceptive measures during study therapy and for at least 3 months after completion of therapy; a negative serum pregnancy test within 72 hours of starting drug is required
* Patients who have a major surgical procedure, or significant traumatic injury within 28 days prior to the first date of treatment on this study, or anticipation of need for major surgical procedure during the course of the study; patients with placement of vascular access device or core biopsy within 7 days prior to the first date of treatment on this study
* Patients with other invasive malignancies, with the exception of non-melanoma skin cancer, who had (or have) any evidence of other cancer present within the last 5 years or whose previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior therapy with this drug

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-04-19 (Actual); Primary Completion 2014-05-01 (Actual); Study Completion 2019-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John K Chan, Principal Investigator — NRG Oncology
Locations (97):
- United States (91):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - University of Colorado Hospital, Aurora, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - AdventHealth Orlando, Orlando, Florida
  - Northside Hospital, Atlanta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Parkland Memorial Hospital, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
- South Korea (6):
  - Keimyung University-Dongsan Medical Center, Jung-Ku, Daegu
  - Samsung Medical Center, Seoul, Korea
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Korea Cancer Center Hospital, Seoul

REFERENCES:
- [Derived] Chan JK, Brady W, Monk BJ, Brown J, Shahin MS, Rose PG, Kim JH, Secord AA, Walker JL, Gershenson DM. A phase II evaluation of sunitinib in the treatment of persistent or recurrent clear cell ovarian carcinoma: An NRG Oncology/Gynecologic Oncology Group Study (GOG-254). Gynecol Oncol. 2018 Aug;150(2):247-252. doi: 10.1016/j.ygyno.2018.05.029. Epub 2018 Jun 18. PMID 29921512

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 4/9/2010 and closed to accrual on 9/30/2013.
Groups:
- SU11248: SU11248 (sunitinib malate) 50 mg per day for 4 weeks followed by 2 weeks off administered in repeated 6-week cycles until disease progression or adverse effects prohibit further therapy
Period: Overall Study
Arm/Group | SU11248
Started | 35
Completed | 30
Not Completed | 5
Not completed — Ineligible - inadequate pathology | 1
Not completed — Ineligible - wrong cell type | 2
Not completed — Refused - Never Treated | 2

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients.
Arm/Group | SU11248
Number analyzed (Participants) | 30
Age, Customized [Number; unit: participants]
  20-29 years | 2
  30-39 years | 1
  40-49 years | 10
  50-59 years | 9
  60-69 years | 7
  70-79 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response Rate (Complete and Partial Response)
Description: Complete and Partial Tumor Response by RECIST 1.1. RECIST 1.1 defines complete response as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm and the disappearance of all non-target lesions and normalization of tumor marker level. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Only those patients who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: CT scan or MRI if used to follow lesion for measurable disease every other cycle for the first 6 months; then every 3 months x 2; then every 6 months thereafter until disease progression for up to 5 years.
Population: Eligible and treated patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | SU11248
Number analyzed (Participants) | 30
percentage of participants | 6.7 [1.2 to 19.5]

2. Primary Outcome: The Percentage of Patients Who Survive Progression Free for at Least 6 Months
Description: Progression-free survival (PFS) was defined as the period from study entry until disease progression, death, or the last date of contact. Progression was based on RECIST 1.1. RECIST 1.1 defines progressive disease as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions or unequivocal progression of non-target lesions is also considered progression.
Time Frame: CT scan or MRI if used to follow lesion for measurable disease every other cycle for the first 6 months
Population: Eligible and treated patients.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | SU11248
Number analyzed (Participants) | 30
percentage of participants | 16.7 [6.8 to 31.9]

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: Every cycle during treatment, then every 3 months for the first 2 years, then every six months for the next three years and then annually, for a total duration of 8.25 years
Population: Eligible and treated patients.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | SU11248
Number analyzed (Participants) | 30
months | 12.8 [6.8 to 17.1]

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the period from study entry until disease progression, death, or the last date of contact. Progression was based on RECIST 1.1
Time Frame: Tumor scans were done every other cycle for the first 6 months; then every 3 months x 2; then every 6 months thereafter for up to 5 years.
Population: Eligible and treated patients.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | SU11248
Number analyzed (Participants) | 30
months | 2.7 [2.5 to 2.9]

5. Secondary Outcome: Number of Participants With Grade 3 or Higher Adverse Events
Description: Grade 3 or higher adverse events were graded by CTC AE v 4.
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment, and up to 5 years in follow-up.
Population: Eligible and treated patients
Measure: Number; unit: participants
Arm/Group | SU11248
Number analyzed (Participants) | 30
participants
  Platelet count decreased | 6
  Anemia | 5
  Fatigue | 4
  Neutrophil count decreased | 4
  Hypertension | 4
  Abdominal pain | 3
  Creatinine increased | 3
  White blood cell decreased | 3
  Nausea | 2
  Vomiting | 2
  Lymphocyte count decreased | 2
  Hypoalbuminemia | 2
  Hyponatremia | 2
  Headache | 2
  Acute kidney injury | 2
  Dyspnea | 2
  Thromboembolic event | 2
  Blood and lymphatic system disorders - other | 1
  Abdominal distension | 1
  Ascites | 1
  Colitis | 1
  Mucositis oral | 1
  Small intestinal obstruction | 1
  Death, NOS | 1
  Edema trunk | 1
  Pain | 1
  Allergic Reaction | 1
  Investigations, other | 1
  Dehydration | 1
  Hyperglycemia | 1
  Neoplasms benign, malignant and unspecified | 1
  Stroke | 1
  Hematuria | 1
  Urinary tract obstruction | 1
  Pleural effusion | 1
  Palmar-plantar erythrodysesthesia syndrome | 1
  Hypotension | 1

6. Other Pre Specified Outcome: Change in Pro-angiogenic Protein Levels
Time Frame: Baseline to up to 5 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Changes in Serum and Plasma Angiogenesis Markers by Enzyme-linked Immunosorbent Assays
Time Frame: Baseline to up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment, and up to 5 years in follow-up.
Arm/Group | SU11248
Serious Adverse Events (participants affected / at risk) | 15/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SU11248 (N=30)
Vomiting (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Pain (General disorders) | 1
Fatigue (General disorders) | 1
Death Nos (General disorders) | 1
Allergic Reaction (Immune system disorders) | 1
Platelet Count Decreased (Investigations) | 2
Creatinine Increased (Investigations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Neoplasms Benign, Malignant And Unspecified (Incl (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Stroke (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic Event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SU11248 (N=30)
Blood And Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 23
Tinnitus (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 5
Hyperthyroidism (Endocrine disorders) | 1
Eye Disorders - Other (Eye disorders) | 1
Flashing Lights (Eye disorders) | 2
Blurred Vision (Eye disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 7
Dry Mouth (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 13
Diarrhea (Gastrointestinal disorders) | 14
Vomiting (Gastrointestinal disorders) | 10
Bloating (Gastrointestinal disorders) | 5
Stomach Pain (Gastrointestinal disorders) | 1
Salivary Duct Inflammation (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Anal Hemorrhage (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 10
Rectal Hemorrhage (Gastrointestinal disorders) | 1
Mucositis Oral (Gastrointestinal disorders) | 14
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 1
Oral Pain (Gastrointestinal disorders) | 2
Abdominal Distension (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 18
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 4
Rectal Pain (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Pain (General disorders) | 3
Localized Edema (General disorders) | 1
Edema Trunk (General disorders) | 3
Edema Limbs (General disorders) | 3
Edema Face (General disorders) | 1
Fatigue (General disorders) | 19
Fever (General disorders) | 2
Chills (General disorders) | 3
Upper Respiratory Infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Investigations - Other (Investigations) | 1
Weight Loss (Investigations) | 1
Platelet Count Decreased (Investigations) | 16
Lymphocyte Count Decreased (Investigations) | 5
Ggt Increased (Investigations) | 1
Creatinine Increased (Investigations) | 3
Neutrophil Count Decreased (Investigations) | 16
White Blood Cell Decreased (Investigations) | 18
Aspartate Aminotransferase Increased (Investigations) | 3
Alkaline Phosphatase Increased (Investigations) | 6
Alanine Aminotransferase Increased (Investigations) | 2
Metabolism And Nutrition Disorders - Other (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 7
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 12
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Peripheral Sensory Neuropathy (Nervous system disorders) | 8
Paresthesia (Nervous system disorders) | 1
Leukoencephalopathy (Nervous system disorders) | 1
Intracranial Hemorrhage (Nervous system disorders) | 1
Headache (Nervous system disorders) | 10
Extrapyramidal Disorder (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 3
Amnesia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 3
Agitation (Psychiatric disorders) | 2
Urinary Urgency (Renal and urinary disorders) | 3
Urinary Tract Obstruction (Renal and urinary disorders) | 2
Urinary Frequency (Renal and urinary disorders) | 1
Renal Calculi (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 5
Hemoglobinuria (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 3
Acute Kidney Injury (Renal and urinary disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 1
Rash Acneiform (Skin and subcutaneous tissue disorders) | 3
Purpura (Skin and subcutaneous tissue disorders) | 1
Periorbital Edema (Skin and subcutaneous tissue disorders) | 1
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 3
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 3
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6
Thromboembolic Event (Vascular disorders) | 3
Hypotension (Vascular disorders) | 2
Hypertension (Vascular disorders) | 10
Hot Flashes (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less